CLINICAL TRIAL: NCT03453437
Title: A Randomized Controlled Trial of a Mindful Self-compassion Intervention to Improve Evaluative Concerns Perfectionism, Depression, Anxiety, and Unhealthy Body Image in College Students
Brief Title: Mindful Self-compassion and Perfectionism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UiBMSC2018
Record Dates: First submitted 2018-01-16; First posted 2018-03-05 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Perfectionism; Depression; Anxiety; Body Image
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Receiving no intervention (control groups will be offered the intervention after the experimental group has completed the course)
- Active group (Experimental): Receiving Mindful Self-Compassion intervention
  Interventions: Behavioral: Mindful Self-Compassion

INTERVENTIONS:
Behavioral: Mindful Self-Compassion — Mindful self-compassion is a course developed by Kristin Neff and Christopher Germer designed to cultivate self-compassion as measured by three subcategories: self-kindness, mindfulness, and a sense of common humanity. This study will shorten the original 8-week course to 5 sessions, and will include interventions and lectures aimed directly toward addressing evaluative concerns perfectionism.
  Arms: Active group

SUMMARY:
The study is a randomized controlled study. A total of 200 students will be invited to participate in a 5-session mindful self-compassion course aimed at increasing self-compassion and reducing maladaptive perfectionism, anxiety, depression, and unhealthy body image. Self-compassion is the ability to show oneself kindness in instances of perceived inadequacy, failure, and suffering by attending to distressing experiences with kindness, mindfulness, and the ability to recognize these as a part of a shared humanity. Twelve participants will be randomly selected for pre- and post interviews to qualitatively evaluate outcome. Ten participants with high perfectionistic tendencies will be selected to participate in a narrative life story interview.

DETAILED DESCRIPTION:
The investigators will test four hypotheses:

1. At baseline, low levels of maladaptive perfectionism, and lower levels of depression, anxiety and body appreciation - reversed, will be related to greater self-compassion. The investigators expect high level of maladaptive perfectionism to be related to lower baseline self-compassion, higher levels of depression and anxiety and lower levels of body appreciation.
2. The intervention, a five session self-compassion intervention, will be sufficient to induce positive changes in perfectionism and psychological symptoms of anxiety, depression and body-appreciation- reversed.
3. Changes in self-compassion will co-vary with changes in maladaptive perfectionism and body appreciation.
4. Higher baseline levels of maladaptive perfectionism will predict greater gains from the intervention, because perfectionistic students will have greater need for a self-compassion intervention.

ELIGIBILITY:
Inclusion Criteria:

* College/university students

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2018-02-03 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
Change in perfectionism | Baseline (two for control group), one week prior to intervention, every week for four weeks until completion of intervention (including one week after last session), 6 months after intervention
  Adaptive perfectionism as measured by the "Personal Standards" subscale and maladaptive perfectionism/evaluative concerns perfectionism as measured by "Doubts about Actions" and "Concern over Mistakes" subscales of the Frost Multidimensional Perfectionism Scale. Personal Standards consists of seven items (6 items for "pure personal standards"), Doubt about Actions consists of four items, and Concern over Mistakes consists of 9 items. All items are on a 5-point Likert scale ranging from strongly disagree to disagree with higher scores indicating most perfectionistic tendencies. Full range: 20-100 with higher scores representing more perfectionistic tendencies. Evaluative concerns perfectionism range: 13-65, higher scores indicate more evaluative concerns perfectionism. Personal standards range: 7-35 with higher scores indicating higher personal standards.

SECONDARY OUTCOMES:
Change in body image | Baseline (two for control group), one week prior to intervention, one week after last session, 6 months after intervention
  Body image as measured by the 13 item Body Appreciation Scale consisting of a 5-point Likert scale. Range: 13-65, lower scores indicating no body appreciation and higher scores indicating greater body appreciation.
Change in depressive tendencies | Baseline (two for control group), one week prior to intervention, every week for four weeks until completion of intervention (including one week after last session), 6 months after intervention
  Depressive tendencies as measured by the 12 item Major Depression Inventory which measures symptoms of depression on a 6-point Likert scale (not at all to all of the time), range: 12-72, with higher scores indicating more symptoms of depression.
Change in anxiety | Baseline (two for control group), one week prior to intervention, every week for four weeks until completion of intervention (including one week after last session), 6 months after intervention
  Anxiety as measured by the 20 item "trait subscale" of the State and Trait Anxiety Inventory. The Inventory consists of a 4-point Likert scale (almost never to almost always), range: 20-80, higher scores indicating greater anxiety.
Change in self-compassion | Baseline (two for control group), one week prior to intervention, every week for four weeks until completion of intervention (including one week after last session), 6 months after intervention
  Assessment of self-compassion with the Self-Compassion Scale short form.Total score range from 12 (no self-compassion) to 60 (high on self-compassion). Higher values represent greater self-compassion, lower scores indicate no self-compassion.

CONTACTS AND LOCATIONS:
Overall Officials: Per-Einar Binder, PhD, Principal Investigator — University of Bergen
Locations (1):
- University of Bergen, Bergen, Hordaland, Norway

REFERENCES:
- [Background] Avalos L, Tylka TL, Wood-Barcalow N. The Body Appreciation Scale: development and psychometric evaluation. Body Image. 2005 Sep;2(3):285-97. doi: 10.1016/j.bodyim.2005.06.002. Epub 2005 Aug 26. PMID 18089195
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Dundas I, Binder PE, Hansen TGB, Stige SH. Does a short self-compassion intervention for students increase healthy self-regulation? A randomized control trial. Scand J Psychol. 2017 Oct;58(5):443-450. doi: 10.1111/sjop.12385. Epub 2017 Aug 28. PMID 28850726
- [Background] Frost, R.O., Marten, P., Lahart, C., Rosenblate R. The dimensions of perfectionism. Cognitive Therapy and Research, 14 (1990), pp. 449-468.
- [Background] Spielberger, C. D., Gorsuch, R. L., Lushene, R., Vagg, P. R., & Jacobs, G. A. (1983). Manual for the State-Trait Anxiety Inventory. Palo Alto, CA: Consulting Psychologists Press.
- [Background] Bech P, Rasmussen NA, Olsen LR, Noerholm V, Abildgaard W. The sensitivity and specificity of the Major Depression Inventory, using the Present State Examination as the index of diagnostic validity. J Affect Disord. 2001 Oct;66(2-3):159-64. doi: 10.1016/s0165-0327(00)00309-8. PMID 11578668
- [Background] Chang, E. C., Linn, N. J., Herringshaw, A. J., Sanna, L. J., Fabian, C. G., Pereraa, M. J., & Marchenkoa, V. V. (2011). Understanding the link between perfectionism and adjustment in college students: Examining the role of maximizing. Personality and Individual Differences, 50(7), 1074.
- [Background] Neff, K. D. (2003). The development and validation of a scale to measure self-compassion. Self and identity, 2(3), 223-250. doi:10.1080/15298860309027
- [Background] Bardone-Cone AM, Sturm K, Lawson MA, Robinson DP, Smith R. Perfectionism across stages of recovery from eating disorders. Int J Eat Disord. 2010 Mar;43(2):139-48. doi: 10.1002/eat.20674. PMID 19308994
- [Background] Boone L, Soenens B, Luyten P. When or why does perfectionism translate into eating disorder pathology? A longitudinal examination of the moderating and mediating role of body dissatisfaction. J Abnorm Psychol. 2014 May;123(2):412-8. doi: 10.1037/a0036254. PMID 24886015
- [Background] Wade TD, Tiggemann M. The role of perfectionism in body dissatisfaction. J Eat Disord. 2013 Jan 22;1:2. doi: 10.1186/2050-2974-1-2. eCollection 2013. PMID 24764525
- [Background] Braun TD, Park CL, Gorin A. Self-compassion, body image, and disordered eating: A review of the literature. Body Image. 2016 Jun;17:117-31. doi: 10.1016/j.bodyim.2016.03.003. Epub 2016 Mar 31. PMID 27038782
- [Background] Breines, J., Toole, A., Tu, C., & Chen, S. (2014). Self-compassion, body image, and self-reported disordered eating. [Journal; Peer Reviewed Journal]. Self and identity, 13(4), 432-448.
- [Background] Kelly AC, Tasca GA. Within-persons predictors of change during eating disorders treatment: An examination of self-compassion, self-criticism, shame, and eating disorder symptoms. Int J Eat Disord. 2016 Jul;49(7):716-22. doi: 10.1002/eat.22527. Epub 2016 Apr 6. PMID 27061929
- [Background] Kelly AC, Vimalakanthan K, Carter JC. Understanding the roles of self-esteem, self-compassion, and fear of self-compassion in eating disorder pathology: an examination of female students and eating disorder patients. Eat Behav. 2014 Aug;15(3):388-91. doi: 10.1016/j.eatbeh.2014.04.008. Epub 2014 May 10. PMID 25064287
- [Background] Pisitsungkagarn K, Taephant N, Attasaranya P. Body image satisfaction and self-esteem in Thai female adolescents: the moderating role of self-compassion. Int J Adolesc Med Health. 2014;26(3):333-8. doi: 10.1515/ijamh-2013-0307. PMID 24114894
- [Background] Albertson, E., Neff, K., & Dill-Shackleford, K. (2015). Self-Compassion and Body Dissatisfaction in Women: A Randomized Controlled Trial of a Brief Meditation Intervention. Mindfulness, 6(3), 444-454. doi:10.1007/s12671-014-0277-3
- [Derived] Woodfin V, Molde H, Dundas I, Binder PE. A Randomized Control Trial of a Brief Self-Compassion Intervention for Perfectionism, Anxiety, Depression, and Body Image. Front Psychol. 2021 Dec 9;12:751294. doi: 10.3389/fpsyg.2021.751294. eCollection 2021. PMID 34955971